CLINICAL TRIAL: NCT04028973
Title: Towards a Better Understanding of Neuromuscular Alterations and Fatigue in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Neuromuscular Fatigue in Chronic Obstructive Pulonary Disease
Acronym: NEUROTIGUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Université de Toulon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-CHITS-03; 2019-A01986-51 (Other: IdRCB by ANSM)
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Neuromuscular fatigue; Muscle; Dual-task; Mental fatigue
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Mental Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Evaluation of fatigue level in BPCO patients (condition 1) (Experimental)
  Interventions: Other: Single then dual task situation
- Evaluation of fatigue level in BPCO patients (condition 2) (Experimental)
  Interventions: Other: Dual then single task situation
- Evaluation of fatigue in control patients (condition 1) (Active Comparator)
  Interventions: Other: Single then dual task situation
- Evaluation of fatigue in control patients (condition 2) (Active Comparator)
  Interventions: Other: Dual then single task situation

INTERVENTIONS:
Other: Single then dual task situation — Firstly, the participants have to perform the fatiguing task in simple task condition (control condition, i.e., muscle contraction alone). Secondly, few days later (between 3 and 7 days later), the participants have to perform the same fatiguing task with a concomitant memory cognitive task (i.e. dual-task condition).
  Arms: Evaluation of fatigue in control patients (condition 1); Evaluation of fatigue level in BPCO patients (condition 1)
Other: Dual then single task situation — Firstly, the participants have to perform the fatiguing task in dual-task condition (i.e. muscle fatiguing contraction with a concomitant memory cognitive task). Secondly, few days later (between 3 and 7 days later), the participants have to perform the same muscle fatiguing task without a concomitant memory cognitive task (i.e. control condition).
  Arms: Evaluation of fatigue in control patients (condition 2); Evaluation of fatigue level in BPCO patients (condition 2)

SUMMARY:
Fatigue is a prevalent symptom in Chronic Obstructive Pulmonary Disease (COPD) that limits patients in their daily living activities. It is now well established that COPD patients may have altered neuromuscular functions compared to healthy individuals. However, the different studies conducted on muscle fatigue in COPD have been done independently of any cognitive solicitation, yet present in most of daily living activities. Therefore, the aim of this research is to evaluate the impact of the disease on neuromuscular fatigue during dual-task situation (simultaneous accomplishment of a muscle contraction and a cognitive task). A better understanding of fatigue in COPD will promote the development of new perspectives in patient management.

The hypothesis is that COPD patients will exhibit increased fatigue level (compared to healthy subjects), particularly during dual-task situation. It is assumed that the higher negative effect associated with the dual-task will be related to different neurophysiological mechanisms (i.e., neuromuscular fatigue, autonomic nervous system activity, mental fatigue).

DETAILED DESCRIPTION:
This study will include three experimental sessions for both COPD patients and healthy participants. These experimental sessions will be performed on three separate days. Each session will last between 1.5 and 2 hours.

The first session will correspond to a familiarization session with the different tests that will be performed during the two next sessions. During this first session, different functional tests will be also performed : 1-minute sit-to-stand tests and postural tests, with and without a concomitant cognitive task.

The second and third sessions will correspond to experimental sessions during which the participants will accomplish a fatiguing task in single or dual-task situation (randomized order). The cognitive task will be a memory cognitive task, called n-back task. The fatiguing tasks will involve submaximal isometric contractions of the knee extensors performed until task failure. The neuromuscular fatigue will be evaluated regularly during the fatiguing tasks (i.e. about each minute) using the magnetic stimulation of the femoral nerve in order to assess to central and peripheral determinants of the neuromuscular fatigue. Moreover, the autonomic nervous system activity (via cardiac recordings), perceived exertion and cognitive performance (in dual-task situation) will be continuously recorded during the fatiguing tasks. Before and after each fatiguing tasks, several questionnaires will be completed (i.e. mood, motivation, subjective workload) in order to evaluate the psychological determinants of performance.

ELIGIBILITY:
Inclusion Criteria:

COPD patients :

* GOLD II - III or IV
* FEV1 <80% of predicted values
* Men and women aged 40 years and over
* French-speaking participant
* BMI <30 kg / m²
* Stable condition (i.e. without exacerbation) for more than 15 days
* Able to express their consent in writing prior to any participation in the study
* Affiliates or beneficiaries of a social security
* Minimum score of 26 on the MMSE questionnaire of 3 months or less

Healthy volunteers :

* Men and women aged 40 years and over
* French-speaking participant
* BMI <30 kg / m²
* No known chronic respiratory, cardiovascular, metabolic, renal or neuromuscular pathologies
* Able to express their consent in writing prior to any participation in the study
* Affiliates or beneficiaries of a social security
* Minimum score of 26 on the MMSE questionnaire of 3 months or less

Exclusion Criteria:

COPD patients :

* Alcoholism, i.e. > 21 glasses a week for men and >14 glasses a week for women
* Psychiatric pathologies or antecedent of behavioral disorders
* Patients treated with oral or systemic corticosteroids (> 0.5 mg / kg / day for > 7 days)
* Contraindication to the application of a magnetic field (i.e. right hip arthroplasty, pelvic / abdominal surgeries)
* Severe vision or hearing problems not corrected
* Patient oxygen dependent
* Patients in exclusion period from another research protocol
* Pregnant women (known pregnancy) or lactating women
* Patient deprived of liberty by a judicial or administrative decision
* Patient subject to a legal protection measure or unable to express their consent
* Patient who is not sufficiently fluent in reading and understanding the French language to be able to consent to participate in the study
* Patient unable to follow study procedures and to respect visits throughout the study period
* Person with a medical history that, in the opinion of the investigator, could interfere with the results of the study
* Any condition that, in the opinion of the investigator, could increase and compromise the safety of the person in the event that he / she participates in the study
* Any other reason that, in the opinion of the investigator, could interfere with the evaluation of the aims of the study

Healthy volunteers:

* Alcoholism, i.e. > 21 glasses a week for men and >14 glasses a week for women
* Psychiatric pathologies or antecedent of behavioral disorders
* Patients treated with oral or systemic corticosteroids (> 0.5 mg / kg / day for > 7 days)
* Contraindication to the application of a magnetic field (i.e. right hip arthroplasty, pelvic / abdominal surgeries)
* Severe vision or hearing problems not corrected
* Subjects in exclusion period from another research protocol
* Pregnant women (known pregnancy) or lactating women
* Regular physical activity with a frequency greater than 3 sessions per week
* Participant deprived of liberty by a judicial or administrative decision
* Participant subject to a legal protection measure or unable to express their consent
* Participant who is not sufficiently fluent in reading and understanding the French language to be able to consent to participate in the study
* Participant unable to follow study procedures and to respect visits throughout the study period
* Person with a medical history that, in the opinion of the investigator, could interfere with the results of the study
* Any condition that, in the opinion of the investigator, could increase and compromise the safety of the person in the event that he / she participates in the study
* Any other reason that, in the opinion of the investigator, could interfere with the evaluation of the aims of the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Endurance time differences between simple and dual-task conditions, in COPD patients compared to healthy participants | 7 days
  The endurance times will correspond to the duration of the fatiguing tasks (simple and dual-task). The endurance time differences between simple and dual-task conditions will be calculated as follows : Endurance time in simple task condition - Endurance time in dual-task condition = Difference of endurance time.

SECONDARY OUTCOMES:
Neuromuscular fatigue of knee extensors | About each minute during the fatiguing tasks lasting about 20 minutes
  The neuromuscular fatigue will be evaluated regularly during the fatiguing tasks using the magnetic stimulation of the femoral nerve , during and after maximal voluntary contraction. Moreover, the muscle activity of the Vastus Lateralis, using non-invasive surface electromyography (sEMG), will be continuously recorded during the fatiguing tasks.
Autonomic nervous system activity | Continuously during the fatiguing tasks lasting about 20 minutes
  Autonomic nervous system activity will be continuously recorded during the fatiguing tasks using cardiac measurements .
Mental fatigue | Continuously during the fatiguing task in dual-task condition, which should last about 20 minutes
  The influence of mental fatigue on the performance will be assessed using the cognitive performance (i.e. rate of correct answers and reaction time) that will be continuously recorded during fatiguing dual-task.
Psychological state | Before, during and after fatiguing task lasting about 20 minutes
  Psychology influence on task performance will be evaluated with questionnaires before, during and after the task. For motivation: 14 items, scores from 0 (not at all) to 4 (extremely), 2 subscales assessing intrinsic and success-based motivation (scores from 0 to 28). For mood: 24 adjectives, scores from 0 (not at all) to 4 (extremely), 6 subscales evaluating fatigue, confusion, vigor, depression, tension and anger (scores from 0 to 16). For Rating-of-Fatigue scale: one score from 0 (not tired) to 10 (exhaustion). For dyspnea: one score from 0 (nothing) to 10 (extremely strong). For Task Load Index: 6 subscales, from 0 (very low) to 20 (very high), measure mental and physical difficulties, time pressure, performance perception, effort perception and frustration. For Sleep Quality Index: 24 questions, 7 subscales from 0 to 3 evaluating subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbance, sleep medication and day dysfunction due to sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc VALLIER, MD PhD, Study Director — Université de Toulon
Locations (2):
- France (2):
  - Université de Toulon, laboratoires LAMHESS et IAPS, La Garde, Var
  - Hôpital d'Instruction des Armées Sainte-Anne, Toulon, Var

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chatain C, Vallier JM, Paleiron N, Cucchietti Waltz F, Ramdani S, Gruet M. Muscle endurance, neuromuscular fatigability, and cognitive control during prolonged dual-task in people with chronic obstructive pulmonary disease: a case-control study. Eur J Appl Physiol. 2025 Feb;125(2):409-428. doi: 10.1007/s00421-024-05608-x. Epub 2024 Sep 21. PMID 39305368